CLINICAL TRIAL: NCT00151021
Title: Automated Step-count Feedback to Promote Physical Activity in Diabetes
Brief Title: Stepping Up to Health: Feedback to Promote Physical Activity in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Michigan Diabetes and Training Center (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: MDRTC 5P60DKK20572
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Pedometer; Behavioral
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Behavior

INTERVENTIONS:
Behavioral: Tailored web-based walking program

SUMMARY:
The primary purpose of this study is to test an Internet based program along with an enhanced pedometer to promote walking in people with diabetes. The major research question to be answered is if counseling and feedback that emphasizes a 10-minute minimum duration for physical activity bouts result in a different pattern of walking behavior compared to counseling and feedback focusing only on total daily accumulated steps.

DETAILED DESCRIPTION:
Objective #1: To develop and test a computer program that automatically collects enhanced pedometer data, records the data in a format suitable for statistical analysis, and generates a personally tailored motivational web page and distributes an e-mail reminder message to encourage the participant to log on to his/her website.

Objective #2: To compare total daily steps in people with diabetes randomized to two different 6-week pedometer and web-based walking interventions. The two interventions will differ only in the emphasis for goal setting and feedback.

Group 1: Emphasizes 10-minute minimum duration of physical activity bouts

Group 2: Emphasizes total daily steps without regard to duration of walking bouts

Objective #3: To compare steps accumulated in walking bouts lasting for at least 10 minutes between the same two groups of participants with diabetes.

Objective #4: To assess the feasibility, cost, dropout rate and participant satisfaction with a pedometer and web-based walking intervention for participants with diabetes.

This study will consist of three phases. Phase I will be the development of a web-based interactive system including data downloading and tailored messages.

Phase II is a usability testing phase in which 8 participants will be recruited to wear the pedometer, interact with the web-based system and give feedback for final development. The Usability phase will occur exactly like the Phase III outlined below except that the participants will be assigned to a study group rather than randomized, and they will be on-study for 2 weeks only - one week for the enrollment phase and one week of the intervention phase. At the end of the intervention week, they will not complete the post survey but will instead complete a feasibility/usability survey and meet with the study staff to help define improvements and adjustments for the Phase III trial. To maximize the Usability Phase, the feedback received from the first four participants will be incorporated in the website before the last four participants are enrolled.

The final phase (Phase III) will include a total of 40 men and women ages > 18 years old, who have Type II Diabetes and are interested in starting a walking program. If they meet eligibility and sign a consent form they will enroll in a randomized control trial comparing two similar interventions to promote walking. Both interventions are 6-week pedometer-based interventions that rely on step-count feedback to motivate participants to increase their walking. Tailored behavioral, informational and motivational messages will be delivered on the website and the enhanced pedometer work by participants will automatically upload time-stamped step count data to a central computer. One of the interventions, the "10 minute bouts" intervention will emphasize bouts of walking lasting at least 10 minutes and of at least moderate intensity. The second intervention called the "total steps" intervention will emphasize total accumulated daily step counts without regard to duration or intensity of walking bouts.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Have type 2 diabetes
* Have a sedentary lifestyle
* Interested in starting a walking program
* Regular computer users who check e-mail at least 5 times a week and have access to a personal computer (PC) with XP or Windows 2000 operating system, 128 MB of memory, and an available universal serial bus (USB) port.
* Can identify a primary care doctor, endocrinologist or cardiologist and obtain written clearance to start a walking program.
* Willing to provide written informed consent
* Can communicate in English

Exclusion Criteria:

* Used a pedometer in past 30 days
* Currently pregnant
* Cannot comfortably walk at least one block
* Cannot obtain written clearance to start a walking program from primary care doctor, endocrinologist or cardiologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-06; Study Completion 2006-01

PRIMARY OUTCOMES:
Step-count bout ratio = 7 day average of steps taken during 10 minute bouts in one day divided by total steps taken during the same day

CONTACTS AND LOCATIONS:
Overall Officials: Caroline R Richardson, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Department of Family Medicine, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Richardson CR, Mehari KS, McIntyre LG, Janney AW, Fortlage LA, Sen A, Strecher VJ, Piette JD. A randomized trial comparing structured and lifestyle goals in an internet-mediated walking program for people with type 2 diabetes. Int J Behav Nutr Phys Act. 2007 Nov 16;4:59. doi: 10.1186/1479-5868-4-59. PMID 18021411